CLINICAL TRIAL: NCT00403169
Title: Phase II Study of CC-5013 in Patients With Advanced Renal Cell Carcinoma (RCC)
Brief Title: Lenalidomide in Treating Patients With Advanced or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-7165; P30CA043703 (NIH); CASE-CCF-7165
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Lenalidomide

ARMS (1):
- Lenalidomide for Advanced RCC (Experimental): 25 mg/day Lenalidomide for 21 days per cycle.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — drug
  Other Names: CC-5013

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of kidney cancer by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well lenalidomide works in treating patients with advanced or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the best response in patients with advanced or unresectable renal cell carcinoma (RCC) treated with lenalidomide.
* Evaluate the response duration, time to tumor progression, and survival of patients with advanced RCC treated with lenalidomide.
* Evaluate the safety of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive oral lenalidomide daily on days 1-21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma (RCC)

  * Advanced or unresectable RCC
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques OR ≥ 10 mm with spiral CT scan
* No brain metastases

  * Brain metastases that have been treated with either radiotherapy or surgery and remain asymptomatic, with no active brain metastases, as shown by CT scan or MRI, for ≥ 6 months are allowed

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if hepatic metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancies within the past 5 years, except for treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, localized prostate cancer, or superficial bladder cancer
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to lenalidomide or thalidomide
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit study compliance
* No hepatitis A, B, or C positivity
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 1 prior systemic therapy for RCC (e.g., chemotherapy, hormonal therapy, immunotherapy)
* At least 4 weeks since prior surgery, radiotherapy, hormonal therapy, chemotherapy, or immunotherapy and recovered
* No prior lenalidomide
* No other concurrent anticancer agents or treatments
* No other concurrent investigational agents
* No concurrent sargramostim (GM-CSF), radiotherapy, or thalidomide

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2004-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Overall response

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States